CLINICAL TRIAL: NCT03884569
Title: Cultivated Limbal Epithelial Transplantation (CLET) for Limbal Stem Cell Deficiency (LSCD): an Observational Study on Safety and Effectiveness
Brief Title: Cultivated Limbal Epithelial Transplantation (CLET) for Limbal Stem Cell Deficiency (LSCD)
Acronym: CLET-4-LSCD
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Citospin (Industry); Red de Terapia Celular (Industry); University of Valladolid (Other)
Responsible Party: Sponsor
Other Study IDs: IOBA201901
Record Dates: First submitted 2019-03-08; First posted 2019-03-21 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Limbal Stem-cell Deficiency
Keywords: limbal stem cell deficiency; corneal failure; limbal epithelial stem cells; ocular surface; corneal blindness
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with CLET: Previously treated with CLET patients are included retrospectively, as the follow-up procedure is already stablished in our centre, and patients treated following standard care or through "drugs-in-special-situation" request in Spain prospectively. Patients are not treated to be included in the study, only the follow-up variables are taken into account.

SUMMARY:
CLET is a published treatment for the management of corneal failure due to extensive LSCD. Due to our previous studies on this novel treatment, the regulatory agency of Spain "Agencia Española de Medicamentos y Productos Sanitarios (AEMPS)" authorized our institution (IOBA-University of Valladolid) to perform this kind of therapy (CLET) in a case-by-case base following the Special Situation Medicines Policy Procedure in Spain. Upon approval of the permanent authorization patients will be included as specified by AEMPS.The objective of this study is to perform a protocolized treatment and follow up so that results can be reported to the scientific community.

ELIGIBILITY:
Total and/or severe LSCD of any etiology in one or both eyes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with corneal failure due to LSCD who accept and sign the informed written consent treatment to be treated with CLET
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Points of improvement in the Single Item Dry Eye Questionnaire (SIDEQ) | 6 months
  The SIDEQ gives a 0-4 score about the presence of dryness, foreign body sensation, burning/stinging, pain, itching, sensitivity to light, and blurred vision, where higher scores indicate higher intensity of the symptom (maximun score: 28). One of the primary outcomes for this work is the improvement in any of the four questionnaires shown here.
Points of improvement about the Ocular Surface Disease Index (OSDI) | 6 months
  The OSDI evaluates ocular surface symptoms with 12 questions, and scores >12 indicate abnormal symptomatology, and >32 means severe symptoms (maximum score 100). One of the primary outcomes for this work is the improvement in any of the four questionnaires shown here.
Points of improvement in the National Eye Institute 25-item Visual Function Questionnaire (NEI-VFQ25) | 6 months
  The visual function-related aspects of the quality of life were evaluated with the NEI-VFQ25, where higher scores on a 0 to 100 scale indicate better function. One of the primary outcomes for this work is the improvement in any of the four questionnaires shown here.
Points of improvement in the Change in Dry Eye Symptoms Questionnaire (CDES-Q) | 6 months
  The CDES-Q evaluates ocular surface symptoms with two questions, CDES-Q1 and CDES-Q2. CDES-Q1 evaluates the change in symptoms occured since the previous examination (same, better or worse). CDES-Q2 evaluates the magnitude of the change in a scale from 0 to 10, where 0 means "slightly better/worse" and 10 means "extremely better/worse". One of the primary outcomes for this work is the improvement in any of the four questionnaires shown here.
Percentage of improvement in corneal conjunctivalization | 6 months
  Percentage of corneal area with conjunctivalization (superficial opacity and/or superficial neovascularization) will be measured.
Complete absence of persistent epithelial defects | 6 months
  Corneal fluorescein staining has to rule out epithelial breakdown

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calonge M, Perez I, Galindo S, Nieto-Miguel T, Lopez-Paniagua M, Fernandez I, Alberca M, Garcia-Sancho J, Sanchez A, Herreras JM. A proof-of-concept clinical trial using mesenchymal stem cells for the treatment of corneal epithelial stem cell deficiency. Transl Res. 2019 Apr;206:18-40. doi: 10.1016/j.trsl.2018.11.003. Epub 2018 Nov 22. PMID 30578758
- [Background] Galindo S, Herreras JM, Lopez-Paniagua M, Rey E, de la Mata A, Plata-Cordero M, Calonge M, Nieto-Miguel T. Therapeutic Effect of Human Adipose Tissue-Derived Mesenchymal Stem Cells in Experimental Corneal Failure Due to Limbal Stem Cell Niche Damage. Stem Cells. 2017 Oct;35(10):2160-2174. doi: 10.1002/stem.2672. Epub 2017 Aug 10. PMID 28758321
- [Background] Lopez-Paniagua M, Nieto-Miguel T, de la Mata A, Galindo S, Herreras JM, Corrales RM, Calonge M. Successful Consecutive Expansion of Limbal Explants Using a Biosafe Culture Medium under Feeder Layer-Free Conditions. Curr Eye Res. 2017 May;42(5):685-695. doi: 10.1080/02713683.2016.1250278. Epub 2016 Dec 2. PMID 27911610
- [Background] Lopez-Paniagua M, Nieto-Miguel T, de la Mata A, Dziasko M, Galindo S, Rey E, Herreras JM, Corrales RM, Daniels JT, Calonge M. Comparison of functional limbal epithelial stem cell isolation methods. Exp Eye Res. 2016 May;146:83-94. doi: 10.1016/j.exer.2015.12.002. Epub 2015 Dec 17. PMID 26704459
- [Background] Ramirez BE, Sanchez A, Herreras JM, Fernandez I, Garcia-Sancho J, Nieto-Miguel T, Calonge M. Stem Cell Therapy for Corneal Epithelium Regeneration following Good Manufacturing and Clinical Procedures. Biomed Res Int. 2015;2015:408495. doi: 10.1155/2015/408495. Epub 2015 Sep 16. PMID 26451369
- [Background] Ramirez BE, Victoria DA, Murillo GM, Herreras JM, Calonge M. In vivo confocal microscopy assessment of the corneoscleral limbal stem cell niche before and after biopsy for cultivated limbal epithelial transplantation to restore corneal epithelium. Histol Histopathol. 2015 Feb;30(2):183-92. doi: 10.14670/HH-30.183. Epub 2014 Jul 30. PMID 25075515
- [Background] de la Mata A, Nieto-Miguel T, Lopez-Paniagua M, Galindo S, Aguilar MR, Garcia-Fernandez L, Gonzalo S, Vazquez B, Roman JS, Corrales RM, Calonge M. Chitosan-gelatin biopolymers as carrier substrata for limbal epithelial stem cells. J Mater Sci Mater Med. 2013 Dec;24(12):2819-29. doi: 10.1007/s10856-013-5013-3. Epub 2013 Jul 28. PMID 23892486
- [Background] Nieto-Miguel T, Galindo S, Reinoso R, Corell A, Martino M, Perez-Simon JA, Calonge M. In vitro simulation of corneal epithelium microenvironment induces a corneal epithelial-like cell phenotype from human adipose tissue mesenchymal stem cells. Curr Eye Res. 2013 Sep;38(9):933-44. doi: 10.3109/02713683.2013.802809. Epub 2013 Jun 14. PMID 23767776
- [Background] Lopez-Paniagua M, Nieto-Miguel T, de la Mata A, Galindo S, Herreras JM, Corrales RM, Calonge M. Consecutive expansion of limbal epithelial stem cells from a single limbal biopsy. Curr Eye Res. 2013 May;38(5):537-49. doi: 10.3109/02713683.2013.767350. Epub 2013 Feb 13. PMID 23405945
- [Background] Nieto-Miguel T, Calonge M, de la Mata A, Lopez-Paniagua M, Galindo S, de la Paz MF, Corrales RM. A comparison of stem cell-related gene expression in the progenitor-rich limbal epithelium and the differentiating central corneal epithelium. Mol Vis. 2011;17:2102-17. Epub 2011 Aug 10. PMID 21850186
- [Background] de la Mata A, Mateos-Timoneda MA, Nieto-Miguel T, Galindo S, Lopez-Paniagua M, Planell JA, Engel E, Calonge M. Poly-l/dl-lactic acid films functionalized with collagen IV as carrier substrata for corneal epithelial stem cells. Colloids Surf B Biointerfaces. 2019 May 1;177:121-129. doi: 10.1016/j.colsurfb.2019.01.054. Epub 2019 Jan 28. PMID 30716697